CLINICAL TRIAL: NCT00450164
Title: Secondary Prophylaxis After Variceal Bleeding: Combined Treatment With Endoscopic Ligation and Nadolol Against Nadolol Associated With Mononitrate of Isosorbide or Prazosin According to Hemodynamic Response.
Brief Title: Secondary Prophylaxis After Variceal Bleeding in Non-Responders
Acronym: KT-2000
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KT-2000
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2007-03-21 (Estimated); Status verified 2007-03

CONDITIONS: Gastrointestinal Hemorrhage; Portal Hypertension; Cirrhosis
Keywords: Variceal bleeding; Secondary profilaxis; Hemodynamic; Portal hypertension
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hypertension, Portal; Fibrosis | interventions — Nadolol; isosorbide-5-mononitrate; Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: esofagic varices ligation
Drug: Nadolol
Drug: Isosorbide mononitrate
Drug: Prazosin

SUMMARY:
Controlled and randomized study comparing combined treatment (nadolol and endoscopic ligation) versus nadolol associated with isosorbide mononitrate or prazosin according to hemodynamic response, in the prevention of esofagic verices rebleeding.

DETAILED DESCRIPTION:
The present is a prospective, randomized, open label study, in parallel groups, in which the patients with hemorrhage caused by esofagic varices will be randomized in two groups of treatment, after control of acute hemorrhage.

All the patients included will receive standard medical treatment with beta - blockers and endoscopic ligation of the esofagic varices.

The control group will be constituted by the patients assigned to receive endoscopic ligation and nadolol (N).

The experimental group will be constituted by patients assigned to receive treatment according to the hemodynamic response.

All patients included in the experimental group will receive pharmacologic treatment with nadolol combined with Isosorbide Mononitrate (MNI) or Prazosin (PZ).

In both groups it will practice a basal hepatic hemodynamic study in the 4th-5th day after their admitance (after achieve hemodynamic stability for at least 48 h and with hemorrhage controlled) and a second control hepatic hemodynamic study 3-4 weeks after the beginning of the pharmacologic treatment, once adjusted doses.

In the experimental group, the responders to N + MNI will keep on this treatment, but nonrespondent in the hemodynamic study will switch treatment to N + PZ and a third hepatic hemodynamic study will be performed 3 to 4 weeks after the dosage adjustement.

The randomization will be stratified according to the degree of hepatic failure measured by Child-Pugh classification (classes A and B versus C) The design is random to avoid bias in the selection of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Any Patient with endoscopically assessed Variceal Bleeding (esofagic and gastric)
* Cirrhosis
* Patient agreement to be included in the study onsentiment signed

Exclusion Criteria:

* Any associated comorbidity with life expectancy lesser than 6 months
* Patient refusement to be included in the study.
* Pregnancy
* Failure to control acute bleeding
* Previous prophylaxis treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2000-11; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Compared efficacy (at least 6 moths of follow-up)

SECONDARY OUTCOMES:
Mortallity
Rebleeding

CONTACTS AND LOCATIONS:
Overall Officials: Candid - Villanueva, Dr., Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Unidad de Sangrantes, HSCSP, Barcelona, Barcelona, Spain